CLINICAL TRIAL: NCT02054312
Title: Phase II Study of Family Based Interpersonal Psychotherapy (FB-IPT) for Depressed Preadolescents
Brief Title: Family Based Interpersonal Psychotherapy (FB-IPT) for Depressed Preadolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Laura Dietz, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH079353
Record Dates: First submitted 2014-02-02; First posted 2014-02-04 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Depressive Disorders
MeSH Terms: conditions — Depressive Disorder | interventions — Person-Centered Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Based Interpersonal Psychotherapy (FB-IPT) (Experimental): Family Based Interpersonal Psychotherapy for Depressed Preadolescents (FB-IPT) is a promising psychosocial treatment for preadolescent depression. It is conceptually rooted in an interpersonal model of depression that focuses on how stress in interpersonal relationships is often related to the onset or maintenance of depressive symptoms. In keeping with adult and adolescent models of IPT, FB-IPT focuses on improving the interpersonal functioning of individuals as a means to improve their depressive symptoms. FB-IPT addresses two domains of interpersonal impairment in depressed preadolescents, parent-child conflict and interpersonal avoidance, and focuses on family relationships, the primary context for children's social and emotional development.
  Interventions: Behavioral: Family Based Interpersonal Psychotherapy (FB-IPT)
- Client Centered Therapy (CCT) (Active Comparator): Child Centered Therapy (CCT), a supportive and nondirective treatment that closely approximates the standard of care for pediatric depression in community mental health. CCT is a manualized treatment for children between the ages of 8-14 based on a Rogerian counseling model. In that model, changes in children's mood and behavior are initiated through their experience of a therapeutic relationship marked by unconditional positive regard, empathic understanding, and therapeutic genuineness.
  Interventions: Behavioral: Client Centered Therapy (CCT)

INTERVENTIONS:
Behavioral: Family Based Interpersonal Psychotherapy (FB-IPT)
  Arms: Family Based Interpersonal Psychotherapy (FB-IPT)
Behavioral: Client Centered Therapy (CCT)
  Arms: Client Centered Therapy (CCT)

SUMMARY:
The investigators proposed a preliminary randomized control trial of Family Based Interpersonal Psychotherapy (FB-IPT), a family-based adaptation of Interpersonal Psychotherapy for Depressed Adolescents (IPT-A; Mufson et al., 2000). Forty-five preadolescent children (ages 8-12) diagnosed with a depressive disorder will be randomized to receive a 14-week course of FB-IPT or Client Centered Therapy (CCT), a supportive nondirective psychotherapy that closely approximates treatment at usual in community mental health clinics. In addition to assessing the feasibility and acceptability of randomization and each of the treatment conditions, this project will evaluate the effects of FB-IPT and CCT across multiple domains, including symptomatology and psychosocial functioning. Preadolescents will be assessed prior to treatment, during treatment (Weeks 3, 7, 11), one week post-treatment, and at 3 and 6 months post-treatment to compare changes in depressive symptoms, global, social, and family functioning. Data on psychosocial risk factors associated with onset and recurrence of preadolescent depression will be collected prior to treatment and at specified intervals post-treatment in order to conduct exploratory analyses on correlates of positive and negative treatment outcomes for Family Based IPT. This data will be used to generate future hypotheses about potential mediators and moderators that will be incorporated into an R01 application for an efficacy study of Family Based IPT.

ELIGIBILITY:
Inclusion Criteria:

* current depressive disorder
* one parent must be willing to participate in treatment

Exclusion Criteria:

* bipolar disorder
* PTSD
* recent abuse
* developmental delay
* autism spectrum disorder

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2010-10; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Childhood Depression Rating Scale -Revised | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laura J Dietz, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute & Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Dietz LJ, Mufson L, Irvine H, Brent DA. Family-based interpersonal psychotherapy for depressed preadolescents: an open-treatment trial. Early Interv Psychiatry. 2008 Aug;2(3):154-61. doi: 10.1111/j.1751-7893.2008.00077.x. PMID 21352148
- [Derived] Dietz LJ, Weinberg RJ, Brent DA, Mufson L. Family-based interpersonal psychotherapy for depressed preadolescents: examining efficacy and potential treatment mechanisms. J Am Acad Child Adolesc Psychiatry. 2015 Mar;54(3):191-9. doi: 10.1016/j.jaac.2014.12.011. Epub 2014 Dec 30. PMID 25721184